CLINICAL TRIAL: NCT01520701
Title: Impact of Applying a Bandage Skin Hydrogel on the Pains of the Head and Neck in Patients With Cancer of Head and Neck Treated With Radiotherapy
Acronym: IPAC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IPAC
Record Dates: First submitted 2012-01-13; First posted 2012-01-30 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; Hydrotac®; radiodermatitis; algia; radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Radiodermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ialuset® application (Active Comparator): Arm with application to the skin Ialuset ® cervical during radiotherapy
  Interventions: Drug: Ialuset®
- bandage skin Hydrosorb (Experimental): Arm bandage skin hydrogel (Hydrotac®) on the skin cervical during radiotherapy
  Interventions: Device: bandage skin Hydrotac®

INTERVENTIONS:
Device: bandage skin Hydrotac® — Patients randomized to the arm with bandage skin will benefit from the application of the bandage skin hydrogel (Hydrotac®) at least 5 hours per day for the duration of treatment (the first day last day of radiotherapy).
  Arms: bandage skin Hydrosorb
Drug: Ialuset® — Patients randomized to receive reference of the application of cervical Ialuset® on skin throughout the treatment period (the first day to last day of radiotherapy).
  Arms: Ialuset® application

SUMMARY:
The investigators hope to get by reduced and delayed acute radiodermatitis following the application of dressings to skin hydrogel Hydrosorb®, a reduction in head and neck pains and improved quality of life of patients with head and neck cancer treated with concomitant radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years old
* Carcinoma oral cavity, pharyngolaryngeal or without lymphadenopathy door
* Patient treated by one of the following diagrams

  * radiotherapy alone
  * postoperative radiotherapy + / - sensitized platinum (cisplatin or carboplatin)
  * ar chemoradiation 5-FU and platinum (the Cetuximab is not allowed)
  * diagram organ preservation (induction chemotherapy and radiotherapy in responders)
* Untreated patients
* Patient should receive conventional radiotherapy or tomotherapy
* Adapted stomatological care
* Life expectancy > 3 months
* WHO score < 2
* Patient stable, not having the time of the examination of evidence of recurrent or progressive malignancy other
* - For patients with an indication of chemotherapy combined with radiotherapy,biological assessments compatible with chemotherapy:

  * WBC > 3000/mm3, Polynuclear > 2000/mm3,Platelets > 150,000/mm3, Creatinine less than 2 times normal; Bilirubin less than 2.5 times normal
* Patient fluent in French
* Affiliation to a system of social security
* Patient has given written consent

Exclusion Criteria:

* Patient with a history of malignancy, outside a basal cell carcinoma or cervical cancer treated and cured
* Patient has at the time of examination signs of recurrence or other neoplasia scalable
* Patient with a history of prior chemotherapy or radiation therapy with the exception of the scheme of organ preservation (induction chemotherapy before radiation)
* For patients with an indication of chemotherapy combined with radiotherapy, contraindication to treatment with specific platinum (cisplatin or carboplatin) with or without 5 Fluorouracil
* Infectious diseases uncontrolled
* Patient is pregnant or lactating or absence of contraception during their reproductive
* Patient hypertensive unbalanced under antihypertensive treatment
* Uncontrolled cardiac disease
* Patients with renal or hepatic
* Known allergy to any component of Ialuset ®
* Patient deprived of liberty under guardianship
* Any medical condition or psychological associate that could compromise the patient's ability to participate in the study
* Inability to undergo medical test for geographical, social or psychological

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2012-02 (Actual); Primary Completion 2022-10 (Actual); Study Completion 2022-10 (Actual)

PRIMARY OUTCOMES:
Impact of applying a bandage hydrogel skin on head and neck pains | end of radiotherapy
  Assessing the impact of applying a bandage hydrogel skin on head and neck pains in patients with cancer of head and neck treated with concomitant radiotherapy by evaluating the proportion of patients with a deterioration in three or more points to their score algia EVA rating scale at the end of treatment compared to that obtained at baseline (D0).

SECONDARY OUTCOMES:
Evaluating the terms of issue of the treatment | during radiotherapy weekly : 1 up to 7 weeks and at 1,3,6,12,18,24,30 and 36 months after radiotherapy
  Evaluating the terms of issue of the treatment (number of interruptions, longer duration of treatment, dose reduction therapeutic influence of psychosocial factors) and quality of life for patients.

CONTACTS AND LOCATIONS:
Overall Officials: David BLANCHARD, MD, Principal Investigator — Centre François Baclesse; Audrey LASNE-CARDON, MD, Principal Investigator — Centre François Baclesse
Locations (7):
- France (7):
  - Centre Maurice TUBIANA, Caen, Calvados
  - CHU, Caen, Calvados
  - Centre François BACLESSE, Caen, Calvados
  - Centre de la Baie, Avranches
  - Clinique Leonard de Vinci, Chambray-lès-Tours
  - centre hospitalier du Cotentin, Cherbourg
  - Centre Guillaume Le Conquérant, Le Havre